CLINICAL TRIAL: NCT06739811
Title: Phoenix: Clinical Evaluation of the Medtronic Implantable Insulin Pump System (MIIPS 2020) in Adult Subjects With Type 1 Diabetes
Brief Title: Clinical Evaluation of the Medtronic Implantable Insulin Pump System (MIIPS 2020) in Adult Subjects With Type 1 Diabetes (CIP347)
Acronym: Phoenix CIP347
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP347
Record Dates: First submitted 2024-12-10; First posted 2024-12-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Type I Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- MIIPS 2020 (Experimental): Subjects implanted with the MIIPS 2020 and treated with intraperitoneal insulin infusion.
  Interventions: Device: Implantable Insulin Pump System

INTERVENTIONS:
Device: Implantable Insulin Pump System — Medtronic Implantable Insulin Pump System (MIIPS 2020)

SUMMARY:
The purpose of this study is to evaluate the clinical performance of the Medtronic Implantable Insulin Pump System (MIIPS 2020) in adult patients with Type 1 diabetes mellitus that cannot be controlled with subcutaneous insulin therapy (including external pump), and presenting with frequent, otherwise unexplained severe hyper- and/or hypoglycemia.

DETAILED DESCRIPTION:
This study is a premarket, interventional, prospective, open-label, multi-center study. It consists of a run-in period, a study period, and a continued access period.

Run-in Period: The purpose of the run-in period is to collect CGM baseline data while subjects are on their current therapy.

Study Period: During the 6-month study period, subjects will be implanted with the MIIPS 2020 and treated with intraperitoneal insulin infusion.

Continued Access Period: Subjects who have completed the entire study period will continue using investigational study devices until those devices are approved for commercial use. Once CE mark is received, the subjects will continue wearing the implanted device.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged ≥ 18 years old.
2. Subject has a clinical diagnosis of type 1 diabetes for ≥ 6 months prior to screening as determined via medical record or source documentation by an individual qualified to make a medical diagnosis.
3. Subject with type 1 diabetes mellitus that cannot be controlled with subcutaneous insulin therapy (including external pump), presenting with frequent, otherwise unexplained severe hyper-and/or hypoglycaemia.
4. Subject has access to a reliable support person, defined as an individual who has daily contact with the subject and knows who to contact in the event of an emergency (i.e., caregiver).
5. Subject has the physical and intellectual ability (in the opinion of the study investigator) to operate the MIIP system and to comply with the data reporting requirements of the study.
6. Subject is willing and able to sign and date informed consent, comply with all study procedures as required during the study.

Exclusion Criteria:

1. Subject is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or device before enrollment into this study, that could impact the outcomes of this study; as per investigator and sponsor judgment.
2. Subject has any other disease or condition that may increase risks during the implant procedure or may preclude the subject from participating in the study, as determined by a physician who is not the principal investigator.
3. Subject has any known or suspected allergy to insulin or implantable materials of the MIIPS (pump and catheter) as determined by a physician.
4. Subject is a woman who is pregnant, of childbearing potential or lactating, and who is neither surgically sterile nor using contraceptives (devices, oral, implanted or other physician-approved contraceptive) at the time of enrollment.
5. Subject is vulnerable, legally incompetent or illiterate.
6. Residence or planned non-pressurized travel at elevations above 10000 feet/3048 meters (commercial airline travel is acceptable).
7. Planning to engage in activities requiring a descent greater than or equal to 10 feet/3 meters below sea level.
8. Subject has an active infection requiring antibiotic treatment.
9. Subject is a person whose body size is not sufficient to accept implantable pump bulk and weight.
10. Subject has a life expectancy of less than 9 months.
11. Subject has diagnosis of illicit drugs abuse disorder.
12. Subject has diagnosis of marijuana abuse disorder.
13. Subject has diagnosis of prescription drugs abuse disorder.
14. Subject has diagnosis of alcohol abuse disorder.
15. Subject who is unwilling or unable to monitor their glucose level or wear a personal continuous glucose monitor.
16. Subject who is unwilling or unable to make programming modifications to the pump based on glucose level readings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Delivery accuracy of MIIPS 2020 | 6 months (4 refill cycles)
  Refill Accuracy= (Total Actual Volume Dispensed)/(Total Theoretical Volume Dispensed)

SECONDARY OUTCOMES:
Refill accuracy at each refill visit | 6 months (4 refill cycles)
  The average of refill accuracy will be summarized at each refill visit
Percentage of pump with accuracy ratio ≤ 85% prompting NaOH rinse | 6 months (4 refill cycles)
  The percentage of pump with refill accuracy ≤ 85%, which prompts NaOH rinse, will be calculated

CONTACTS AND LOCATIONS:
Locations (3):
- France (2):
  - Centre Hospitalier Universitaire De Montpellier, Montpellier, France
  - Hôpital Européen Marseille, Marseille
- Isala Zwolle, Zwolle, Netherlands, Netherlands

IPD SHARING:
Plan to Share IPD: No